CLINICAL TRIAL: NCT06644911
Title: The Effect of Maternal Obesity on Umbilical and Uterine Artery Doppler in Term Pregnancy : a Cross-sectional Study
Brief Title: Obesity Doppler in Term Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Professor, Assiut University
Other Study IDs: Doppler-150
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Doppler Measurement of Uterine Artery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal weight pregnant women: Normal weight (body mass index 18.5-24.9 kg/m2)
- Obese pregnant women: women (body mass index ≥ 30 kg/m2)

SUMMARY:
Maternal obesity is an epidemic in the developed world like Egypt. There are many pregnancy-associated complications including pre-eclampsia, gestational diabetes, and increased rates of septic wound after cesarean delivery. As a potential explanation of the etiology of complications due to maternal obesity, the role of endothelial dysfunction in the systemic and peripheral vasculatures has been hypothesized. It has been proposed that some adverse pregnancy outcomes in obese patients may be mediated by placental insufficiency. Utero-placental insufficiency is typically associated with fetal growth restriction and low birth weight.

Umbilical and uterine artery Doppler is widely accepted as a useful tool for monitoring high-risk pregnancies.

Normally, uterine artery vascular impedance gradually decreases until the late mid-trimester, owing to the establishment of a low-resistance placental circulation. Obesity has little impact on uterine vascular changes reflected by the early uterine artery PI. However, in the second trimester, extreme obesity appears to impair the normal continued drop in uterine vascular resistance. Many studies have examined the relationship between BMI and Doppler changes in high-risk pregnancies, but few have addressed these changes in low-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. Gestational age ≥ 37 weeks
3. Absence of fetal structural abnormalities
4. Absence of maternal comorbidities and/or complications.
5. Obese women (BMI ≥ 30 kg/m2) [11].
6. Normal weight (BMI 18.5-24.9) [11].

Exclusion Criteria:

1. Placenta previa
2. Women with antepartum hemorrhage.
3. Smokers and alcohol consumers
4. Preeclampsia
5. Diabetes mellitus
6. Women need urgent termination of pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The difference between uterine and umbilical artery Doppler resistant index | at 37 weeks of pregnancy
  The difference between uterine and umbilical artery Doppler indices between normal weight and obese pregnant women ≥ 37 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes